CLINICAL TRIAL: NCT01619410
Title: Asymptomatic Colonization With S. Aureus After Therapy With Linezolid or Clindamycin for Acute S. Aureus Skin and Skin Structure Infections in Patients With Comorbid Conditions: A Randomized Trial
Brief Title: Asymptomatic Colonization With S. Aureus After Therapy With Linezolid or Clindamycin for Acute Skin Infections
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow accrual
Sponsor: University of Chicago (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-0550
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Results first posted 2019-07-24 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-10

CONDITIONS: Skin Diseases, Bacterial; Abscess
MeSH Terms: conditions — Skin Diseases, Bacterial; Abscess | interventions — Linezolid; Clindamycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- linezolid (Active Comparator)
  Interventions: Biological: Linezolid
- Clindamycin (Active Comparator)
  Interventions: Biological: Clindamycin

INTERVENTIONS:
Biological: Linezolid — Linezolid 600 mg every 12 hours for 7 days
  Arms: linezolid
Biological: Clindamycin — Clindamycin 300 mg po every 6 hours for 7 days
  Arms: Clindamycin

SUMMARY:
In this pilot study, the objective is to determine the prevalence of asymptomatic carriage of S. aureus in patients with ABSSSIs and minor cutaneous abscesses after therapy with either linezolid or clindamycin at 40 days after the completion of therapy. Secondarily, the investigators will assess the efficacy of linezolid vs. clindamycin in the empiric therapy of ABSSSIs and minor cutaneous abscesses, as well as the genotypic spectrum of S. aureus isolates causing ABSSSIs or minor cutaneous abscesses and colonization in the target patient population before and after therapy. Given the results of a recent study on linezolid and vancomycin and the investigator's own experience, it is hypothesized that persistent MRSA carriage will be less common after therapy with linezolid for ABSSSIs and minor cutaneous abscesses than it is with oral clindamycin.

ELIGIBILITY:
Inclusion Criteria:

* having an ABSSSI or a minor cutaneous abscess treated in the ED
* age 18 years or older
* any one or more of the following co-morbidities:

  * diagnosis of diabetes mellitus
  * obesity with a BMI >35
  * chronic kidney disease
  * coronary artery disease
  * peripheral vascular disease

Exclusion Criteria:

* known history of or current thrombocytopenia
* Currently taking anti-depression medication
* Current or recent hospitalization
* Known current alcohol or drug abuse
* Known or suspected hypersensitivity to any ingredient of the study drugs
* Irregular heart rate and blood pressure measurements
* Fevers or low body temperature
* Known psychiatric condition
* Superficial skin infection
* Skin infection caused from an animal bite
* Recent treatment with antibacterials
* Pregnancy

Other protocol related inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Z David, MD, PhD, Principal Investigator — University of Chicago
Locations (2):
- United States (2):
  - Grady Memorial Hospital, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Linezolid | Clindamycin
Started | 14 | 11
Completed | 7 | 7
Not Completed | 7 | 4
Not completed — Lost to Follow-up | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Linezolid | Clindamycin | Total
Number analyzed (Participants) | 14 | 11 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (15.4) | 40.5 (11.9) | 42.0 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 7 | 1 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 11 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 11 | 24
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 11 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Presence of Staphylococcus Aureus After Treatment With Linezolid Versus Clindamycin
Description: Asymptomatic carriage of Staphylococcus aureus at the 40-day visit will be compared in the patients assigned to receive linezolid to the patients assigned to receive clindamycin.
Time Frame: 40 days after completion of treatment
Population: Only subjects returning for the 40-day outcome measurement were included in this analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Linezolid | Clindamycin
Number analyzed (Participants) | 7 | 7
Participants | 3 | 2
Statistical Analysis 1: Comparison: Linezolid vs Clindamycin; Test type: Superiority; p = 1.0, Fisher Exact

2. Secondary Outcome: Number of Participants With Clinical Response of Skin Infections to Treatment -- 7 Days
Description: The efficacy of linezolid versus clindamycin in the treatment of skin infections will be measured using treatment outcomes of cure, treatment failure, or relapse.
Time Frame: 7 days after completion of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Linezolid | Clindamycin
Number analyzed (Participants) | 10 | 7
Participants
  Cure | 10 | 7
  Treatment failure | 0 | 0
  Relapse | 0 | 0

3. Secondary Outcome: Number of Participants With Clinical Response of Skin Infections to Treatment -- 40 Days
Description: as for outcome 2
Time Frame: 40 days after completion of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Linezolid | Clindamycin
Number analyzed (Participants) | 9 | 7
Participants
  Cure | 9 | 6
  Treatment failure | 0 | 0
  Relapse | 0 | 1

4. Secondary Outcome: The Type of of Staphylococcus Aureus Present at the Diagnosis Will be Compared to the Type of Staphylococcus Aureus Present After Treatment
Description: The genotype of Staphylococcus aureus which is found to be the cause of the skin infection will be be compared to the genotype of Staphylococcus aureus present after treatment. Comparisons will will be made between the linezolid and clindamycin treatment groups.
Time Frame: 40 days after completion of treatment
Population: No data available due to samples being lost as a result of equipment issues.
Arm/Group | Linezolid | Clindamycin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 40 days
Arm/Group | Linezolid | Clindamycin
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/11
Other Adverse Events (participants affected / at risk) | 0/14 | 0/11

LIMITATIONS AND CAVEATS:
The anticipated enrollment of 152 subjects wasn't achieved. There was slower accrual because the epidemiology of S. aureus infections changed & fewer eligible patients presented. Thus, the study is underpowered for the primary outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No